CLINICAL TRIAL: NCT05108948
Title: Research of Factors Determining the Improvement of Quality of Life at One Year of Adult Patients Treated for Spinal Deformity : Observational Study (COFTASD)
Brief Title: Research of Factors Determining the Improvement of Quality of Life at One Year of Adult Patients Treated for Spinal Deformity (COFTASD)
Acronym: COFTASD
Status: Recruiting | Type: Observational
Sponsor: Elsan (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A01753-38
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Spinal Deformity
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spinal deformity operated patients
  Interventions: Behavioral: Quality of life questionnaires; Procedure: Radiography

INTERVENTIONS:
Behavioral: Quality of life questionnaires — Oswestry Disability Index Scoliosis Research Society-22R Short Form 36 Health Survey Questionnaire Tobacco, Alcohol, Prescription medication, and other Substance use Core Outcome Measures Index : back and neck
Procedure: Radiography — Spinal radiography : full, face, profile

SUMMARY:
The objective of this study is to find the predictive factors of improvement of the quality of life of operated patients from spinal deformity.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years-old
* Diagnosis of Adult Spinal Deformity with any of the deformity characteristics following:

  * Scoliosis with a Cobb angle ≥ 20 °
  * Vertical sagittal axis (SVA) ≥ 5 cm
  * Pelvic tilt ≥25 °,
  * Thoracic kyphosis with a Cobb angle ≥ 60 °
* Eligible for surgery
* Having given their participation agreement
* Affiliate or beneficiary of a social security scheme

Exclusion Criteria:

* Age under 18 years-old
* Patient unlikely to comply with follow-up
* Patient with long-term complete paraplegia
* Patient unable to understand and answer questionnaires in due to language difficulties or cognitive impairment
* Pregnant or breastfeeding woman
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient over 18 years-old with spinal deformity operated
Sampling Method: Non-Probability Sample
Enrollment: 866 (Estimated)
Dates: Start 2021-10-23 (Actual); Primary Completion 2031-10-23 (Estimated); Study Completion 2041-10-23 (Estimated)

PRIMARY OUTCOMES:
Factors associated with improved oswestry disability score | 15 years
  The factors associated with an improvement in the ODI score, 1 year after surgery, will be sought among the initial characteristics (before surgery) and within 3 months after surgery. An improvement in ODI score is defined as a decrease in score at 1 year of at least 10 points from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique du dos, Bruges, France